CLINICAL TRIAL: NCT04904536
Title: An International, Investigator Initiated and Conducted, Pragmatic Clinical Trial to Determine Whether 40mg Atorvastatin Daily Can Improve Neurocognitive Function in Adults With Long COVID Neurological Symptoms
Brief Title: Statin TReatment for COVID-19 to Optimise NeuroloGical recovERy
Acronym: STRONGER
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: University of Sydney (Other); Monash University (Other); The Alfred (Other); Universidad del Desarrollo (Other); Chinese University of Hong Kong (Other); Clinica Alemana de Santiago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X21-0113
Record Dates: First submitted 2021-05-21; First posted 2021-05-27 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Neurocognitive Impairment, Mild
Keywords: clinical trial; COVID-19; neurological symptoms; atorvastatin
MeSH Terms: conditions — Lymphoma, Follicular; COVID-19; Neurologic Manifestations | interventions — Atorvastatin; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Medication Arm (Experimental): 6-monthly supplies of atorvastatin 40mg on top of standard care for a period of 12 months.
  Interventions: Drug: Atorvastatin
- Standard Care Arm (Active Comparator): Standard care for a period of 12 months.
  Interventions: Other: Standard Care

INTERVENTIONS:
Drug: Atorvastatin — 40mg atorvastatin + standard care daily for 12 months.Atorvastatin 40mg has TGA approval for general marketing for the treatment of hypercholesterolaemia and cardiovascular prevention under a number of manufacturer names.The study medication selected will be the atorvastatin 40mg (Apotex) which is scored, and allows down-titration to 20mg should a participant develop symptoms.The study medication will be packaged, labelled and dispensed directly to particpants by the Syntro Health pharmacy in Australia. A comparable atorvastatin 40mg is being sourced in Chile, and will be dispensed from the pharmacy of the Clínica Alemana de Santiago. Similarly, a comparable atorvastatin 40mg is being sourced in Hong Kong, and will be dispensed from the site's pharmacy.
  Arms: Study Medication Arm
Other: Standard Care — Standard care for neurological symptoms as a result of COVID-19 infection.
  Arms: Standard Care Arm

SUMMARY:
STRONGER is an international, investigator initiated and conducted, pragmatic clinical trial to determine whether 40mg atorvastatin daily can improve neurocognitive function in adults with long COVID neurological symptoms. The objective is to determine effectiveness of treatment with 40mg atorvastatin over 12 months on attenuating cognitive decline and neuroinflammatory biomarkers in adults with long COVID neurological symptoms. The study design is a prospective, randomised, open-label, blinded endpoint (PROBE) study of atorvastatin 40mg on top of standard care, in patients with long COVID neurological symptoms.

DETAILED DESCRIPTION:
Question: Does treatment with 40mg atorvastatin over 12 months attenuate cognitive decline and neuroinflammatory biomarkers in adults with long COVID neurological symptoms? Aims: In 410 adults who report ongoing alteration of their memory, thinking, concentration or mood after COVID-19 diagnosis, this pragmatic clinical trial aims to determine the effects of standard-dose atorvastatin on improving neurological outcomes with sensitive measures of cognitive function and brain MRI.

Outcome measures include; Primary - processing speed, assessed on the oral Symbol Digit Modalities Test (SDMT). Key Secondary - white matter free water measured on diffusion MRI brain imaging. Other - other components of cognitive function; other health assessments; other MRI markers of cerebral white matter integrity, iron load, cerebral perfusion, and glutathione for oxidative stress; cost-effectiveness compared to standard care. The study sites are established at centralised research clinics located at: The Brain and Mind Centre of the University of Sydney; Alfred Medical Centre linked to Monash University, a research clinic associated with Clínica Alemana Universidad del Desarrollo, Santiago, Chile, and a research clinic associated with The Chinese University of Hong Kong. Additional sites may be set up as required.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* History of COVID-19 that is confirmed by a positive polymerase-chain-reaction (PCR) test,rapid antigen test (RAT) or as per the state guidelines for COVID-19 diagnosis at the time of screening
* Any ongoing neurological symptoms as a result of COVID-19 (e.g. problems with memory, concentration, sleep disturbance and fatigue) that are identified through administration of the checklist of symptoms on the Somatic and Psychological Health Report (SPHERE) questionnaire, or reported loss of smell (anosmia)
* Able to fully participate in all procedures, including cognitive assessments
* Able and willing to provide written informed consent

Exclusion Criteria:

* Evidence of dementia and/or significant cognitive impairment on screening (i.e: Blind Montreal Cognitive Assessment [MoCA] score <19/22 in conjunction with clinical assessment)
* Severe co-morbid medical or psychiatric condition that prevents participation
* History of traumatic brain injury with loss of consciousness (>30 mins) within the last 2 years
* Ongoing long-term use for a clear indication (e.g. secondary cardiovascular prevention in high-risk individuals) or any contraindication (e.g. previous adverse reaction) of statin use
* Evidence of severe or significant liver disease, defined as any of the following: acute viral hepatitis; chronic active hepatitis; chronic active hepatitis; cirrhosis; or elevated biochemical function markers i.e. ALT or AST >3x the ULN or eGFR <30mL/min/1.73m2
* Creatine kinase (CK) levels > 2x upper limit of normal (ULN)
* Female of child-bearing potential that is unable or unwilling to use reliable method of contraception, breastfeeding, or planning a pregnancy
* For a sub-group of participants undergoing MRI - any contraindication to MRI due to metallic body parts or claustrophobia
* Medical history of a disorder that might, in the opinion of the attending clinician, put the participant at significant risk if they were to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Neurological Recovery | 12 months
  Processing speed, assessed on the oral Symbol Digit Modalities Test (SDMT)

SECONDARY OUTCOMES:
Brain Imaging | 12 months
  White matter free water measured on diffusion MRI brain imaging

CONTACTS AND LOCATIONS:
Overall Officials: Craig Anderson, MD, Principal Investigator — The George Institute
Locations (1):
- The George Institute for Global Health, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Delfino C, Carcel C, Lin X, Munoz-Venturelli P, Naismith SL, Woodward M, Peters R, Wijesuriya N, Law M, Harding IH, Wang X, Elliott J, Leder K, Hutchings O, Stecher X, Zoungas S, Anderson CS. STatin TReatment for COVID-19 to Optimise NeuroloGical recovERy (STRONGER): study protocol for a randomised, open label clinical trial in patients with persistent neurological symptoms after COVID-19 infection. BMJ Open. 2025 Apr 14;15(4):e089382. doi: 10.1136/bmjopen-2024-089382. PMID 40228860

DOCUMENTS (1):
  • Study Protocol (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT04904536/Prot_000.pdf